CLINICAL TRIAL: NCT05946993
Title: Linking In With Advice and Supports for Men Impacted by Metastatic Cancer
Acronym: LIAM Mc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Irish Cancer Society (Other); Cancer Research@UCC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 22052
Record Dates: First submitted 2023-05-10; First posted 2023-07-14 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Survivorship; Prostate Cancer; Kidney Cancer; Urothelial Tract/Bladder Cancer, Nos; Testicular Cancer; Penile Cancer
Keywords: cancer; prostate; survivorship
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms; Urologic Neoplasms; Testicular Neoplasms; Penile Neoplasms; Neoplasms | interventions — Physical Therapy Modalities; Psychiatric Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Other): Participants will attend 12-week programme that will include twice weekly exercise and assessment sessions.
  Interventions: Other: Physiotherapy; Other: Dietitian Support; Other: Nursing and Psychosocial

INTERVENTIONS:
Other: Physiotherapy — participant will have 2 x 1h exercise classes per week with a physiotherapist, who will develop individualized plans based on medical history and scan reviews. Participants will be progressively guided through the programme, incrementally increasing in intensity or with modifications based on symptomatic presentation. This will be based on their baseline strength and cardiovascular fitness testing and grounded on evidence-based protocols previously demonstrating an effect in this patient population. Individualised tailored exercise programme which includes strength and conditioning.
Other: Dietitian Support — The main goal of the nutritional intervention is to improve the diet quality of each patient using a standardized nutrition assessment, offering evidence-based diet group education and developing personalized nutrition goals. Participants will be progressively guided through the nutrition education programme; with modifications to the individual's usual diet, thereby recognizing personal eating patterns and preferences, which form the basis for individualized dietary counselling. The dietary counselling identifies the type, amount, and frequency of feeding and specifies the caloric/protein level to attain, together with any restrictions and limited or increased individual dietary components.
Other: Nursing and Psychosocial — Nursing, Psycho-oncology, pastoral care and social work-led sessions to inform participants on items including diagnosis shock, acceptance, coping with relationship changes with their partner and their roles, fear of uncertainty and the future, medication management, masculinity (male values being strong, capable, independent), practical management of bills, and household tasks. There will be an inclusion of practical information sessions including health systems information and managing side effects such as urinary symptoms, hot flushes, penile shortening, and loss of body hair.

SUMMARY:
To evaluate the feasibility of introducing a men's cancer survivorship programme into routine follow up care in patients with advanced genitourinary malignancies.

DETAILED DESCRIPTION:
Study design: Sequential Cohorts/ Parallel Sampling Groups Specific Aim: To assess the feasibility of a comprehensive multidisciplinary interventional programme for men living with advanced/metastatic genitourinary cancers Sample size: 72

Entry criteria: Advanced / metastatic genitourinary cancer (including prostate, kidney, urothelial tract, testicular and/or penile cancers), provided they meet the following conditions:

* Prostate cancer - Histologically confirmed prostate cancer and must have commenced Androgen Deprivation Therapy (ADT) in the form of a gonadotropin-releasing hormone (GnRH) analogue or a GnRH receptor antagonist and/or an androgen receptor antagonist and/or undergone bilateral orchidectomy for prostate cancer.
* Urothelial tract cancer - Stage II - IV urothelial tract cancer after completion of primary treatment with systemic therapy
* Kidney cancer - Stage II - III renal cell cancer
* Testicular cancer - Stage II - III testicular cancer after completion of primary treatment
* Penile cancer - • Stage III - IV penile cancer after completion of primary treatment with systemic therapy
* Currently on active surveillance (i.e. no active systemic therapies at present) or continuing on maintenance systemic therapy, provided they do not have ongoing adverse events which will impact their participation at the time of commencing the 12-week intervention.
* Note: Men with resected disease (adjuvant setting) are eligible if they have commenced or completed adjuvant systemic therapy within the past 12 months and have recovered from these treatments at the time of commencing the 12-week programme from ongoing systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged ≥ 18 years of age at the time of study enrolment.
2. Willing to participate in a 12-week intervention programme and follow up procedures as outlined in the Schedule of Activities section.
3. ECOG performance status 0-2.
4. Recovery to CTCAE Grade ≤2 adverse events from all prior therapies, or adequately recovered adverse events whereby, whereby the PI feels they will not impact the participants ability to complete the 12-week intervention.
5. Disease-specific inclusion criteria:

   Prostate cancer:
   * Histologically confirmed prostate cancer
   * Must have commenced Androgen Deprivation Therapy (ADT) in the form of a gonadotropin-releasing hormone (GnRH) analogue or a GnRH receptor antagonist and/or an androgen receptor antagonist and/or undergone bilateral orchidectomy for prostate cancer. Men must have received last ADT treatment within 12 months of starting the programme or have ongoing treatment-related side effects at the time of commencing the programme if ADT has been discontinued due to toxicity.
   * Patients without histologically confirmed cancer are eligible if both the treating physician and the study PI agree that the patient's history is unambiguously indicative of advanced prostate cancer (e.g. high Prostate-specific antigen (PSA) responsive to ADT in prostate cancer).

   Urothelial tract cancer:
   * Stage II - IV urothelial tract cancer (muscle-invasive, node positive or metastatic disease) after completion of primary treatment with systemic therapy (including in the neoadjuvant or adjuvant setting) and/or surgery and recovery from these treatments to a satisfactory level.
   * Patients with metastatic disease continuing on maintenance systemic therapy are permitted if they do not have ongoing CTCAE Grade >2 adverse events which will impact their participation at the time of commencing the 12-week programme.

   Kidney cancer:

   • Stage II - III renal cell cancer (clear cell or non-clear cell histologies permitted) after nephrectomy who required and have commenced or completed adjuvant systemic therapy within the past 12 months and have recovered from these treatments to CTCAE Grade ≤2 or do not have ongoing CTCAE Grade >2 adverse events at the time of commencing the 12-week programme from ongoing systemic therapy.

   Or

   • Stage IV renal cell cancer (clear cell or non-clear cell histologies permitted) where the participants are continuing on stable dose of maintenance systemic therapy and do not have ongoing CTCAE Grade >2 adverse events at the time of commencing the 12-week programme.

   Testicular cancer:

   • Stage II-III testicular cancer after completion of primary treatment with systemic therapy and/or surgery within the past 12 months and recovery of all adverse events from these treatments to CTCAE Grade ≤2.

   Penile Cancer:
   * Stage III - IV penile cancer (node positive, recurrent or metastatic disease) after completion of primary treatment with systemic therapy (including in the neoadjuvant or adjuvant setting) and/or surgery and recovery from these treatments to CTCAE Grade ≤2.
   * Patients with metastatic disease continuing maintenance systemic therapy are permitted if they do not have ongoing CTCAE Grade >2 adverse events which will impact their participation at the time of commencing the 12-week programme.
6. Participation in other translational or interventional clinical trials is permitted provided the above disease-specific inclusion criteria are met.
7. Signed consent form by the participant or a legally authorized representative (LAR).

Exclusion Criteria:

1. Persons who, in the opinion of the researcher or supervising clinician, are unable to cooperate adequately with the study protocol, for example those receiving systemic therapy for a concurrent cancer diagnosis, those with organ system dysfunction which would impact their safe participation in the study, or other uncontrolled medical illness that would impact their safe participation in the study.
2. Recent (within 12 months) participation in a study/programme involving a lifestyle intervention (e.g diet, exercise, survivorship).

   1. Note: Per discretion of PI as to whether may impact the outcome of this study intervention.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by a purposefully designed feasibility questionnaire | At week 12
  The feasibility of introducing a men's cancer survivorship programme into routine follow up care in patients with advanced genitourinary cancer. Purposefully designed feasibility questionnaire will be used. All scores will be linearly transformed to a 0 to 100 scale.
Feasibility as assessed by a purposefully designed feasibility questionnaire | At 6-month post intervention timepoint
  The feasibility of introducing a men's cancer survivorship programme into routine follow up care in patients with advanced genitourinary cancer. Purposefully designed feasibility questionnaire will be used. All scores will be linearly transformed to a 0 to 100 scale.
The acceptability of introducing a men's cancer survivorship programme into routine follow up care in patients with advanced genitourinary cancer | At week 12
  Purposefully designed feasibility questionnaire will be used. All scores will be linearly transformed to a 0 to 100 scale.
The acceptability of introducing a men's cancer survivorship programme into routine follow up care in patients with advanced genitourinary cancer | At the 6-month post intervention timepoint
  Purposefully designed feasibility questionnaire will be used. All scores will be linearly transformed to a 0 to 100 scale.

SECONDARY OUTCOMES:
Change from Baseline in Health related-Quality of Life Questionnaire (QLQ) scores assessed by European Organization for the Research and Treatment of Cancer (EORTC) | Baseline and at the end of the 12-week programme
  Quality of Life survey; European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QoL).
  All patients will answer at the baseline and at the end of the intervention EORTC QLQ-C30 (30 items). The scoring will be performed according to the EORTC scoring manual. All scores will be linearly transformed to a 0 to 100 scale.
Change from Baseline in Fatigue related-Quality of Life Questionnaire (QLQ) scores | Baseline and at the end of the 12-week programme
  Cancer related fatigue score; European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-FA12).
  All patients will answer at the baseline and at the end of the intervention, week 12. All scores will be linearly transformed to a 0 to 100 scale.
Change from Baseline in weight. | Baseline and the programme endpoint (12 weeks).
  The dietitian will perform physical assessments of each patient at the baseline and at the end of the study. The dietitian will record the weight in kg.
Change from Baseline in muscle strength and mass. | Baseline and the programme endpoint (12 weeks).
  The physiotherapist will perform physical assessments of each patient at the baseline and at the end of the study. The physiotherapist will measure the muscle strength and mass through leg extension and biceps curl in kg.
Change from Baseline in 6-minute walk test. | Baseline and the programme endpoint (12 weeks).
  The physiotherapist will perform 6-minute walk test and measure it in metres (m).
Change from Baseline in muscle strength scores on handgrip measurements | Baseline and the programme endpoint (12 weeks).
  The dietitian will perform physical assessments to each patient at the baseline and at the end of the study. Muscle strength will be measured using hand grip strength (HGS) based on the Jamar Dynamometer (Model 091011725).
Change from Baseline in Diet intake scores from multiple 24-hour recalls, complemented by a Food Frequency Questionnaire (FFQ) | Baseline and the programme endpoint (12 weeks).
  All patients will answer at the baseline and at the end of the intervention the FFQ. All patients will answer at the baseline and at the end of the intervention the Food Frequency Questionnaire. Data will be entered in to the FFQ European Prospective Investigation into Cancer and Nutrition (EPIC) Tool for Analysis (FETA). FETA calculates the average daily intake of 46 nutrients and 14 food groups, for each individual. The default nutrients list provides a description of each nutrient/food group and the units used. The nutrient data for the FFQ foods have come from McCance and Widdowson's "The Composition of Foods (5th edition)" and its associated supplements.
Change from Baseline in Diet quality scores from The World Cancer Research Fund/American Institute for Cancer Research (WCRF/AICR) standardised scoring system (Shams-White et al 2019). | Baseline and the programme endpoint (12 weeks).
  All patients will answer at the baseline and at the end of the intervention the WCRF/AICR. The higher the score, the better Diet quality.
Change from Baseline in BMI scores. | Baseline and the programme endpoint (12 weeks).
  The dietitian will perform physical assessments of each patient at the baseline and at the end of the study. Weight and height will be combined to report BMI in kg/m^2. Weight will be reported in kg.
Change from Baseline in Lean Body Mass (LBM) scores. | Baseline and the programme endpoint (12 weeks).
  The dietitian will perform physical assessments of each patient at the baseline and at the end of the study. Weight and body fat will be combined to report LBM in kg*(Percentage body/100).
Change from Baseline in waist circumference scores. | Baseline and the programme endpoint (12 weeks).
  The dietitian will perform physical assessments of each patient at the baseline and at the end of the study. Waist circumference will be measured in cm.
Change from Baseline in Segmental Body Composition scores assessed measured by Body Composition Monitor bioimpedance spectroscopy (BIS). | Baseline and the programme endpoint (12 weeks).
  The dietitian will perform physical assessments on each patient at the baseline and at the end of the study. Weight (Kg) and body fat (%) and Total Body Water (TBW) will be combined to report the Body Composition score.
Change from Baseline in Nutritional risk scores assessed by the Malnutrition Screening Tool (MST) | Baseline and the programme endpoint (12 weeks).
  All patients will complete the MST at the baseline and at the end of the intervention. The higher the score, the higher risk of malnutrition.
Self-care agency and its relationship to quality of life and symptoms experienced | Baseline and the programme endpoint (12 weeks).
  * Instruments to measure self-care agency include the ASAS-R
  * Additional Assessments as identified by the scoping review will be included in the Expansion Phase. The higher the score, the better the self-care agency.
The resource utilisation of signposted services among participants in the 12-week intervention programme | Baseline and the programme endpoint (12 weeks). A high score represents high functionality problems.
  Quality-adjusted life-year (QALY) (EQ-5D-5L). A high score represents high functionality problems.
Satisfaction of participants and Health Care Professionals with the programme and their perceptions of the systems usability. | At the programme endpoint (12 weeks)
  Qualitative analysis of Usability, Satisfaction and Feasibility Questionnaire Participants, health care professionals and the broader team involved in the development and implementation of the programme will be invited to provide feedback after the completion of their involvement in the study. The higher the score, the better usability and satisfaction from the participant

CONTACTS AND LOCATIONS:
Overall Officials: Jack Gleeson, MB, Principal Investigator — Cork University Hospital
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noonan B, Bredin P, Cahill AM, Corkery S, Johnston KE, Medved K, Cusack AM, Hegarty J, Saab MM, Cushen SJ, Connolly R, Palmer B, Dahly D, Murphy M, Bambury RM, Gleeson JP. Study protocol: LIAM Mc trial (Linking In with Advice and supports for Men impacted by Metastatic cancer). PLoS One. 2025 Apr 3;20(4):e0313454. doi: 10.1371/journal.pone.0313454. eCollection 2025. PMID 40179061